CLINICAL TRIAL: NCT00002215
Title: A Randomized, Double-Blind Study of MKC-442 Combined With Viracept in Patients Who Are Epivir + Retrovir Experienced and Are Protease Inhibitor- and Non-Nucleoside Reverse Transcriptase Inhibitor-Naive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 292A; MKC-303
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; Reverse Transcriptase Inhibitors; Viral Load; Nelfinavir; Uracil
MeSH Terms: conditions — HIV Infections | interventions — emivirine; Nelfinavir

INTERVENTIONS:
Drug: Emivirine
Drug: Nelfinavir mesylate

SUMMARY:
To compare the proportion of patients whose plasma HIV-1 RNA level falls and remains below the limit of quantification by the Roche Amplicor Monitor (400 copies/ml)[AS PER AMENDMENT 8/4/98: 50 copies/ml] between weeks 0 and 24. To determine the short-term safety and tolerability of MKC-442 plus nelfinavir (Viracept) plus dual nucleoside analogs. To determine the time to viral failure and time to tolerability failure through Week 48 of therapy.

DETAILED DESCRIPTION:
In this randomized, placebo-controlled study, patients are allowed to switch at entry to d4T plus 3TC or d4T plus ddI based on investigator and patient preference. Patients are stratified based on the number of nucleoside reverse transcriptase inhibitor (NRTI) treatments that are changed at entry and on screening HIV-1 RNA (obtained within 30 days of entry) as follows: switched 1 NRTI and 10,000-50,000 copies/ml vs switched 1 NRTI and greater than 50,000 copies/ml vs switched 2 NRTIs and 10,000-50,000 copies/ml vs switched 2 NRTIs and greater than 50,000 copies/ml. Patients are randomized within each of these strata to 1 of the following treatment arms:

Arm 1: MKC-442 placebo plus nelfinavir. Arm 2: MKC-442 plus nelfinavir. Arm 3: MKC-442 plus nelfinavir (higher dose). Treatment is administered for 48 weeks. Patients who are considered virologic successes at Week 48 may continue to receive MKC-442 at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

At least 1 different nucleoside analog, e.g., 3TC, d4T, or ddI (excluding zidovudine).

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia.
* Short courses (less than 21 days) of acyclovir for acute treatment.
* Recombinant erythropoietin or G-CSF for Grade 3 or greater anemia and neutropenia, respectively.
* Allowed only with caution and close patient monitoring:
* Ketoconazole, fluconazole, itraconazole, and grapefruit juice.
* Medications metabolized by cytochrome P450.
* Oral contraceptives, contraceptive implants such as Norplant, or injection-type contraceptives such as Depo-Provera only if not sole method of contraception.

Patients may have:

* HIV-1 RNA greater than 10,000.
* No active AIDS-defining illnesses.
* Prior experience with 2 nucleoside analogues and able to switch to at least 1 different non-nucleoside analog, e.g., lamivudine (3TC), stavudine (d4T), or didanosine (ddI) with HIV-1 RNA 10,000 copies/ml or less. [AS PER:
* 8/4/98 AMENDMENT].
* [AS PER AMENDMENT 8/4/98:
* Nucleoside analog-naive patients must have HIV-1 RNA greater than 50,000 copies/ml.].

Prior Medication:

Allowed:

Treatment with 2 nucleoside analogs. Note:

* able to switch to at least 1 different nucleoside analog e.g., lamivudine (3TC), stavudine (d4T), or didanosine (ddI), while on study [AS PER AMENDMENT 8/4/98].

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active AIDS-defining illnesses.
* Malabsorption syndrome or severe chronic diarrhea within 30 days of entry, or inability to consume adequate oral intake due to chronic nausea, emesis, or abdominal or esophageal discomfort. [AS PER AMENDMENT 8/4/98].
* Inadequately controlled seizure disorder [AS PER AMENDMENT 8/4/98].
* Any intercurrent illness that could affect viral load determination [AS PER AMENDMENT 8/4/98].

Concurrent Medication:

Excluded:

* Zidovudine.
* Immunomodulators (e.g., systemic corticosteroids, interleukin-2, or interferons). [AS PER AMENDMENT 8/4/98].
* Rifampin, rifabutin, phenobarbital, and hydantoin.
* Amiodarone, quinidine, astemizole, terfenadine, ergot derivatives, midazolam, triazolam, and cisapride.
* Neurotoxic agents (e.g., vincristine, thalidomide). [AS PER AMENDMENT 8/4/98].

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* History of > grade 2 peripheral neuropathy.
* Patients with an acute and clinically significant medical event within 30 days of screening.

Prior Medication:

Excluded:

* Protease inhibitors.
* Non-nucleoside reverse transcriptase inhibitors.

Excluded within 30 days of study drug administration:

* Immunomodulators (e.g., systemic corticosteroids, interleukin-2, or interferons). [AS PER AMENDMENT 8/4/98].
* Rifampin, rifabutin, phenobarbital, and hydantoin.
* Amiodarone, quinidine, astemizole, terfenadine, ergot derivatives, midazolam, triazolam, and cisapride.
* Immunotherapeutic vaccines.
* Cytotoxic chemotherapeutic agents [AS PER AMENDMENT 8/4/98].

Prior Treatment:

Excluded within 30 days of study drug administration:

Radiation therapy [AS PER AMENDMENT 8/4/98].

Risk Behavior:

Excluded:

Current alcohol or illicit drug use that, in the opinion of the investigator, may interfere with ability of patient to comply with dosing schedule and protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anderson Clinical Research, Pittsburgh, Pennsylvania, United States